CLINICAL TRIAL: NCT05838547
Title: PET-MR Imaging of Natriuretic Peptide Receptor C (NPR-C) in Carotid Atherosclerosis With Cu[64]-25%-CANF-Comb-II
Brief Title: CANF-Comb-II PET-MR in Atherosclerosis Multisite
Status: Recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: Cedars-Sinai Medical Center (Other); University of California, Santa Barbara (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Pamela Woodard, MD, HM Wilson Professor of Radiology, Washington University School of Medicine
Other Study IDs: 202210116; 123,617 (Other: Food and Drug Administration (FDA) eIND Number); R01HL159803 (NIH)
Record Dates: First submitted 2023-04-09; First posted 2023-05-01 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Carotid Atherosclerosis; Asymptomatic Carotid Artery Stenosis; Carotid Artery Atheroma
Keywords: Stroke; TIA; Vascular Disease; Cardiovascular Disease
MeSH Terms: conditions — Carotid Artery Diseases; Stroke; Vascular Diseases; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Carotid plaque tissue specimens will be collected at the time of surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients treated with Optimal Medical Therapy (OMT) alone.: Asymptomatic carotid artery stenosis (ACAS) patients with known carotid artery atherosclerosis by ultrasound/Doppler or other carotid imaging ≥ 60% diameter stenosis who are clinically referred for OMT alone.
  Interventions: Drug: 64Cu-25%-CANF-Comb
- Patients treated with OMT and carotid endarterectomy (CEA).: Asymptomatic carotid artery stenosis (ACAS) patients with known carotid artery atherosclerosis by ultrasound/Doppler or other carotid imaging ≥ 60% diameter stenosis who are clinically referred for OMT and CEA.
  Interventions: Drug: 64Cu-25%-CANF-Comb

INTERVENTIONS:
Drug: 64Cu-25%-CANF-Comb — Patients treated with OMT alone that are not treated with CEA will receive an intravenous injection of 4-6 mCi of 64Cu-25%-CANF-Comb radiotracer for PET/MR imaging at the initial imaging visit and at 12-18 months, or earlier if they develop symptoms. While 12-18 months is the preferred window for repeat imaging, if imaging during this time frame is not achievable, the patient may return anytime throughout the remainder of the study.
  Groups: Patients treated with Optimal Medical Therapy (OMT) alone.
Drug: 64Cu-25%-CANF-Comb — Patients treated with OMT and CEA will receive an intravenous injection of 4-6 mCi of 64Cu-25%-CANF-Comb radiotracer for PET/MR imaging at the initial imaging visit.
  Groups: Patients treated with OMT and carotid endarterectomy (CEA).

SUMMARY:
The goal of this observational study is to learn more about plaque biology in asymptomatic carotid artery stenosis (ACAS) patients through imaging. The main questions it aims to answer are:

* To determine the ability of 64Cu-CANF-Comb positron emission tomography (PET) to risk stratify ACAS patients for stroke event, to include transient ischemic attack or remote ipsilateral intervention.
* To further understand the role of Natriuretic Peptide Receptor C (NPRC) in the evolution of carotid atherosclerosis.

Participants will be asked to undergo a carotid PET-magnetic resonance imaging (MRI) examination to assess whether the carotid atherosclerosis uptake of 64Cu-CANF-Comb as measured by PET-MRI correlates with patient outcomes (stroke, transient ischemic attack, or remote ipsilateral intervention).

DETAILED DESCRIPTION:
This is an NIH-funded, Phase II, multicenter, open-label patient outcomes imaging study. Patients will undergo carotid PET/MRI after intravenous injection of 4-6 milliCuries (mCi) of the FDA Exploratory Investigational New Drug (eIND)-approved nanoparticle PET radiotracer (64Cu-C-type atrial natriuretic factor (CANF)-Comb). A total of 80 subjects will be recruited to this study. These subjects will be asymptomatic carotid artery stenosis (ACAS) patients with known carotid artery atherosclerosis by ultrasound/Doppler or other carotid imaging ≥ 60% diameter stenosis. These patients will be asked to undergo a carotid PET/MRI at a single time point 12-24 hours after intravenous injection of the 64Cu-CANF-Comb radiotracer.

Based on promising results from a proof of concept study, the investigators have devised an imaging protocol to determine the ability of 64Cu-25%-CANF-Comb PET to risk stratify ACAS patients treated with optimal medical therapy (OMT) alone with respect to patient outcomes. In this observational study, 80 patients with ACAS ≥ 60% will undergo 64Cu-25%-CANF-Comb PET/MRI. Patients will be maintained on either OMT alone or receive OMT and carotid endarterectomy (CEA) as determined by their treating vascular surgeon prior to imaging.

A total of 80 subjects, both men and women (≥18 years of age), will be recruited at Washington University (WU) and Cedars Sinai, with approximately 59 patients recruited at WU and approximately 21 patients recruited at Cedars Sinai. Patients will be asked to undergo carotid PET/MRI after intravenous injection of 64Cu-25%-CANF-Comb. These 80 subjects will be asymptomatic carotid artery stenosis (ACAS) patients with known carotid artery atherosclerosis by ultrasound/Doppler or other carotid imaging ≥ 60% diameter stenosis. These patients will be asked to undergo a carotid PET/MRI at a single time point 12-24 hours after intravenous injection of the 64Cu-25%-CANF-Comb radiotracer. Patients treated with OMT alone will undergo repeat PET/MRI at 12-18 months, or earlier if they develop symptoms. While 12-18 months is the preferred window for repeat PET/MRI, if imaging during this time frame is not achievable, the patient may return anytime throughout the remainder of the study. PET/MRI changes over time will be used to further understand the biology of carotid plaque evolution after treatment with OMT.

At the time of imaging, the investigators will record baseline medications to include any antiplatelet, statin, anti-hypertension, and diabetes medications (OMT), and basic risk factors and demographic information (e.g. diabetic, hypertensive, smoker, hypercholesterolemia), in addition to the patient's age and sex. Vital signs, a blood draw, and urinalysis will be obtained at baseline and at time of imaging (12-24 hrs after injection). A physical examination will be obtained at baseline and at the time of imaging. Telephone follow-up will occur within 48-72 hours (2-3 days) after discharge and then every 3 months (+/- 5 days) until the end of the study to assess for ipsilateral ischemic cerebrovascular event (TIA, stroke) or remote ipsilateral carotid intervention. This outcomes data will be used to answer the primary objective of this project.

ELIGIBILITY:
Inclusion Criteria:

* Adults, 18 years of age or older
* Asymptomatic carotid artery stenosis patients who have undergone carotid Doppler/ultrasound imaging or other carotid imaging which have demonstrated a ≥ 60% diameter carotid artery stenosis.
* The treating surgeon has planned either treatment with optimal medical therapy (OMT) alone, or OMT and carotid endarterectomy (CEA) surgical intervention.

Exclusion Criteria:

* Inability to receive and sign informed consent.
* Patients with an unstable clinical condition that in the opinion of the Sponsor-Investigator or designee precludes participation in the study.
* Inability to tolerate up to 60 minutes in a supine position with arms down at sides for PET-MR imaging.
* Prior history of CEA or carotid artery stent procedure on the ipsilateral side.
* Past medical history of TIA or stroke within the last 6 months.
* Unwilling to comply with study procedures and/or unable to be available for the duration of the study outlined in the protocol.
* Contraindications to MR imaging (pacemaker, brain aneurysm clips, shrapnel, claustrophobia, etc.).
* Currently pregnant or lactating. All female subjects of childbearing potential must have a documented negative pregnancy test (serum or urine hCG) performed within 24 hours immediately prior to the administration of 64Cu-25%-CANF-Comb or documented post- menopausal defined as the cessation of menses for ≥ 12 months or documentation of having a bilateral oophorectomy and/or hysterectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals ≥18 years of age with asymptomatic carotid artery stenosis.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of patients reporting ipsilateral ischemic cerebrovascular event (TIA, stroke) or remote ipsilateral carotid intervention | Through study completion, up to 4 years.
  Patients will be contacted every 3 months after PET/MR imaging to assess for interval ipsilateral ischemic cerebrovascular event. In patients treated with OMT, it is anticipated that higher 64Cu-CANF-Comb PET signal (SUV) will correlate with increased ipsilateral ischemic cerebrovascular event (TIA, stroke) or remote ipsilateral carotid intervention (CEA surgery or stent placement); PET signal (SUV) will be assessed as a marker of risk for event in comparison to anatomic features of vulnerable plaque on MRI, with the goal of determining 64Cu-CANF-Comb PET signal above which suggests ACAS at higher risk.

SECONDARY OUTCOMES:
Changes in 64Cu-CANF-Comb PET signal - OMT | 12-18 months (preferred); through study completion, up to 4 years.
  Patients treated with OMT will be imaged at baseline and at 12-18 months, or earlier if they develop symptoms, to determine interval change in 64Cu-CANF-Comb PET signal (SUV) over time. While 12-18 months is the preferred window for repeat imaging, if imaging during this time frame is not achievable, the patient may return anytime throughout the remainder of the study.
PET signal relative to presence of targeted receptor, NPR-C and histopathological features of plaque vulnerability - CEA surgery as Treatment | Immediately after surgery.
  In patients who initially undergo CEA, PET signal (SUV) will be compared to ex vivo plaque vulnerability and NPRC cellular distribution to facilitate understanding of gene expression using immunohistochemistry (IHC) and cell lineage/origin through single cell RNA (scRNA)/cellular indexing of transcriptomes and epitopes (CITE)-seq.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Woodard, MD, Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - Cedars Sinai Medical Center, Los Angeles, California
  - Washington University in St. Louis, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No